CLINICAL TRIAL: NCT06663371
Title: The Impact of Integrated Neuromuscular Training Intervention on the Basic Physical Fitness of Military Personnel
Brief Title: The Impact of IntegBasic Physical Fitness Rated Neuromuscular Training Intervention on the of Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Liu (Other)
Responsible Party: Sponsor-Investigator, Yang Liu, Doctor, Wuhan Sports University
Organization: Wuhan Sports University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Basic Physical Fitness
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Chronic Ankle Instability,CA; Basic Physical Fitness
Keywords: Integrated Neuromuscular Training; Military Population; Basic Physical Fitness
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: There is no specific relevant model to refer to for use.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Neuromuscular Training (Experimental): Integrative Neuromuscular Training (INT) is an interdisciplinary training paradigm that amalgamates cutting-edge concepts and practices from the realms of athletic training, physical therapy, biomechanics, and neuroscience. The genesis of INT dates back to the late twentieth century to the early twenty-first century, a period marked by a burgeoning understanding of motor control and neuromuscular coordination. Experts in the fields of sports science and rehabilitation began to explore a training modality designed to holistically enhance athletic performance while concurrently reducing the risk of injury.
  The central tenet of INT is to optimize the coordination of the neuromuscular system and the synergistic action among muscle groups, thereby deepening functional movement training and integrating specific training components. These components include, but are not limited to, strength, balance, velocity, agility, fatigue resistance, and plyometric training. This methodology is not sol
  Interventions: Behavioral: Basic Physical Fitness
- Traditional Physical Training (Placebo Comparator): Traditional Physical Training (TPT) involves a set of exercises with limited variation and fixed movement paths, conducted under stable conditions. This method primarily enhances muscle strength and endurance but often falls short in integrating with specific sports requirements and developing athletes' specialized skills.TPT emphasizes basic athletic attributes like strength, speed, and flexibility, which are vital for competition. Yet, it tends to focus on bulking up muscles and isolating body parts, potentially leading to higher injury risks and suboptimal performance.The concept of TPT is conservative, drawing on traditional sports training without fully embracing modern sports science and rehabilitation. However, as our understanding of motor control and neuromuscular coordination advances, modern training is becoming more holistic and scientific, prioritizing specialized movements, balance, and multi-joint coordination to boost the effectiveness of strength training.
  Interventions: Behavioral: Traditional Physical Training

INTERVENTIONS:
Behavioral: Basic Physical Fitness — The single module training paradigm followed a circuit-style format, with each training module consisting of 6 to 8 distinct exercise movements. Taking the INT training intervention on Mondays as an example, the training protocol involved completing one major module (e.g., plyometric exercises) before transitioning to another module (e.g., core stability exercises). Specific exercise methods, such as box jumps, were performed until all sets were completed before moving on to the next exercise (e.g., continuous depth jumps).
  Other Names: Speed; Strength; Balance; Agility
  Arms: Integrated Neuromuscular Training
Behavioral: Traditional Physical Training — In the fundamental strength training, a circuit training modality is employed, with each training segment comprising 5 to 7 exercise movements. For instance, a series of squat exercises is performed initially, followed by upper body strength training such as bench presses; each movement must be completed with the specified number of sets and repetitions before proceeding to the next exercise. Explosiveness training enhances the rapid contraction capabilities of the muscles through a series of jumping and throwing movements, while flexibility exercises improve the range of motion of muscles and joints through a combination of static and dynamic stretching.
  Other Names: Speed; Strength
  Arms: Traditional Physical Training

SUMMARY:
Objective: The study aims to evaluate the efficacy of an 8-week integrated neuromuscular training intervention on the fundamental physical fitness parameters of military personnel, encompassing strength, velocity, agility, and equilibrium.

Methodology: The research randomly allocated 20 military students from the National University of Defense Technology into two cohorts, utilizing an experimental methodology with longitudinal assessments at the onset, midpoint, and conclusion of the intervention to quantitatively assess the influence of the integrated neuromuscular training on velocity and agility. Participants in both the experimental and control groups were evaluated one week prior to the intervention, at the fourth week, and one week post-intervention. Statistical analysis involved a two-factor repeated measures ANOVA to compare measures across the three time points, while paired-sample t-tests were applied for pre-post comparisons. The experimental group engaged in an 8-week integrated neuromuscular training regimen, consisting of three 90-minute sessions per week, culminating in a total of 24 sessions. Concurrently, the control group adhered to a conventional physical training schedule, also structured around three 90-minute sessions per week, over the same 24-session period, thereby ensuring parity in total training duration and frequency between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-24 years old
* Students with corresponding military status
* Meeting the diagnostic criteria for functional movement screen assessment
* No history of psychological or psychiatric disorders, and not participating in other physical training during the experimental period
* Capable of cooperating to complete the corresponding training and testing, and will not withdraw from the experiment without cause

Exclusion Criteria:

* Major sports injuries within the past 2 years, including fractures, ligament tears, muscle or tendon ruptures, and recurrent dislocations of joints
* Patients with cardiovascular and cerebrovascular diseases and related internal organ conditions
* Failure to pass the functional movement screen test
* Individuals with injuries or discomfort in other areas

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Vertical-Jump Test | 8 weeks
  Vertical-Jump Test: The testing equipment used is the Swiss Myotest explosiveness testing device. Before the start of the test, participants completed familiarization exercises, jogging, stretching, and other routine warm-up activities. The best score out of three attempts was recorded. According to previous research, the test-retest reliability of the vertical jump test under the experimental conditions of this study is 0.993.
Balance Test | 8 weeks
  Balance Test: The Y-balance test (YBT) was used for measurement, following the testing patterns from studies by Plisky et al. and Xu Fei et al. . Specifically, the participant stands on the Y-balance test device with one leg, barefoot, and the other leg's foot is used to slowly push the test board to the furthest distance in three directions: anterior (A), posteromedial (PM), and posterolateral (PL). The sequence is first with the right leg supporting and then with the left leg supporting. Each direction is measured three times, and the maximum distance is taken for analysis. During the test, participants are required to keep their feet stationary and their hands off the anterior superior iliac spine. After the test, the composite score of the YBT for both legs is calculated based on the distances in the three directions for both the left and right legs, which is used to evaluate the participant's balance ability. The calculation formula is [(A + PM + PL) / (3 × lower limb leng
Maximum Strength (1RM, 1 Repetition Maximum) | 8 weeks
  Maximum Strength (1RM, 1 Repetition Maximum): Before the official test, participants are required to perform familiarization exercises without weights, adhering to the standard techniques for the squat and bench press movements. Subsequently, an indirect test for maximum strength is conducted . The calculation formula by Brzycki et al. for 1RM is used: 1RM = weight repeated / (1.0278 - 0.0278 × number of repetitions). For the squat test, participants are instructed to maintain a fixed foot stance and toe angle, with heels always in contact with the ground, and the thighs should be parallel to or slightly below the ground level during each squat, with knees not extending beyond the toes . For the bench press test, participants are required to ensure that the barbell touches the chest before pressing the arms upward until they are fully extended. Research by Kravitz et al. indicates that the 1RM test has a high degree of accuracy.
100m Sprint Test | 8 weeks
  100m Sprint Test: Participants undergo two trials of the 100m sprint test. Prior to the official test, they all engage in 20 minutes of regular warm-up activities, including light jogging and stretching. They are instructed to use a standing start and to exert their maximum effort; upon hearing the start signal, they begin running. There is a 10-minute rest period between the two trials. The test is timed by professional referees with a precision of 0.01 seconds. To ensure consistency, the best performance out of the two trials is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Changsha, China

IPD SHARING:
Plan to Share IPD: No
It involves personal privacy.

REFERENCES:
- [Derived] Liu P, Liu Y, Hao X, Cheng N, Kang J, Xiao Z, He P, Yan J. The impact of an 8-week integrated neuromuscular training on strength, speed, and agility in military personnel: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 May 22;17(1):127. doi: 10.1186/s13102-025-01172-9. PMID 40405304